CLINICAL TRIAL: NCT03814694
Title: Cut Down on Carbohydrate Usage in the Diet of Type 2 Diabetes; Mechanisms of Effective Therapy of Diabetes by Selective Choice of Macronutrients. The Hypo-energetic Study.
Brief Title: Cut Down on Carbohydrate Usage in the Diet of Type 2 Diabetes. The Hypo-energetic Study
Acronym: CutDM-Hypo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: University of Copenhagen (Other); University of Aarhus (Other); The Danish Dairy Research Foundation, Denmark (Other); Arla Foods (Industry)
Responsible Party: Principal Investigator, Mads N Thomsen, Principal Investigator, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CUTDM-HYPO
Record Dates: First submitted 2019-01-08; First posted 2019-01-24 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Diabetes Mellitus, Type 2; Overweight and Obesity
Keywords: Weight Loss; Diet, Carbohydrate-Restricted; Diet, High-Protein; Insulin Resistance; Non-alcoholic Fatty Liver Disease; Metabolic Syndrome
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity; Weight Loss; Insulin Resistance; Non-alcoholic Fatty Liver Disease; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRHP Diet (Experimental): Hypo-energetic carbohydrate-reduced high-protein (CRHP) dietary intervention with a controlled 5-7% loss in body weight.
  Interventions: Dietary Supplement: CRHP Diet
- CD Diet (Active Comparator): Hypo-energetic conventional diabetes (CD) dietary intervention with a controlled 5-7% loss in body weight.
  Interventions: Dietary Supplement: CD Diet

INTERVENTIONS:
Dietary Supplement: CRHP Diet — Dietary macronutrient composition of 30 E% from carbohydrate, 30 E% from protein and 40 E% from fat
  Arms: CRHP Diet
Dietary Supplement: CD Diet — Dietary macronutrient composition of 50 E% from carbohydrate, 17 E% from protein and 33 E% from fat
  Arms: CD Diet

SUMMARY:
Scientific evidence for the dietary treatment of type 2 diabetes (T2D) is insufficient, which is why the investigators aim to reform dietary recommendation to the overweight or obese patient with type 2 diabetes. This clinical study will examine the effect of a highly controlled hypo-energetic carbohydrate-reduced high-protein (CRHP) diet intervention under caloric restriction-induced body weight loss as a treatment modality in T2D. The investigators hypothesize that this intervention compared to the conventional diabetes (CD) diet with similar loss in body weight improves metabolic control and cardiovascular risk profile in T2D by:

* Reducing diurnal and postprandial glycaemia, thereby facilitating a significant reduction in HbA1c
* Reducing ectopic lipid deposits in liver, muscle and pancreas
* Improving lipid profile towards a less atherogenic profile
* Improving metabolic actions of insulin, through increased sensitivity and β-cell function
* Reducing diurnal blood pressure with no adverse effect on heart rate variability

DETAILED DESCRIPTION:
The present study will be performed as a 6-week randomized fully controlled feeding study, which will address the effect of the hypo-energetic CRHP diet compared with the hypo-energetic CD diet with the macronutrient composition currently recommended to patients with T2D combined with a caloric restriction-induced 5-7% body weight loss on T2D. The study includes n=80 T2D patients.

Measurements include fasting blood samples every 2 weeks during the 6 weeks of the study. Additionally, larger measurement programs will be undertaken at baseline and after 6 weeks, including MRi/s for liver, pancreas and muscle fat content and visceral and subcutaneous adipose tissue; DXA scans for body composition; oral glucose tolerance tests (OGTT); continuous glucose monitoring (CGM); diurnal blood pressure and holter recording. Questionnaires of health-related quality of life, level of physical activity and satiety by visual analogue scale will be performed at baseline and week 6 as well as fecal and diurnal urine sampling.

To ensure a similar body weight loss between intervention groups as well as participants, aimed at 5-7%, caloric intake during the 6 weeks of the study will be hypo-energetic adjusted for each participant according to estimated daily total energy expenditure (TEE). A calculation requiring sex, age, weight and height will be performed to estimate resting energy expenditure (REE), which multiplied with the participant's physical activity level (PAL) will estimate TEE, and thus with an initial caloric deficit of 5% determine the caloric content in the hypo-energetic diet for each participant. Additionally, participants will be weighed twice a week and caloric content adjusted accordingly to ensure a controlled body weight loss.

It is important to recognize that the CRHP diet and the CD diet principally do not differ in the quality of carbohydrate and protein. Thus, this study is unable to address a potential benefit of changes in quality of carbohydrate; however, both diet interventions exhibit a relatively low glycemic index of maximum 55.

Until week 6 diets will be prepared and distributed from the research kitchen of the Department of Nutrition, Exercise and Sports, Faculty of Science, University of Copenhagen, Denmark, to optimize compliance and adherence to the prescribed diet. Following this period and again after approximately 3 months participants will be invited to group sessions with dietician guidance on how to sustain their body weight loss and continue with their assigned diet. A follow-up visit at week 30 will include a blood sample, a spot urine sample and body weight measurement.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes with HbA1c between 48 mmol/mol and 97 mmol/mol with or without metformin and dipeptidyl peptidase-4 (DPP-4) inhibitors
* Overweight or obesity with BMI ≥ 25 kg/m2 and desired weight loss
* Non-smokers for > 1 year
* Willingness to abstain from alcohol for 6 weeks
* Hemoglobin > 7 mmol/L for men and > 6 mmol/L for women
* Estimated glomerular filtration rate (eGFR) > 30 mL/min/1.73 m2

Exclusion Criteria:

* Critical illness as evaluated by the principal investigator
* Systemic corticosteroid treatment, e.g. prednisolone
* Reported or journalized severe food allergy or intolerance
* Reported or journalized severe gut disease e.g. Crohn's disease, Coeliac disease etc.
* Reported or journalized alcohol dependence syndrome
* Injectable diabetes medication, including insulin and GLP-1 analogues
* Sulfonylureas (SUs) and sodium-glucose cotransporter 2 (SGLT-2) inhibitors, unless discontinuation is possible, in which case a 2-month wash-out is mandatory
* Repeated fasting plasma glucose > 13.3 mmol/L
* Urine albumin / creatinine ratio > 300 mg/g
* Lactation, pregnancy or planning of pregnancy during the study
* Inability, physically or mentally, to comply with the procedures required by the study protocol, as evaluated by the principal investigator
* Presently participating in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2020-07-22 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Change in glycated hemoglobin (HbA1c) during 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  The change in HbA1c will be assessed during 6 weeks of fully provisioned hypo-energetic CRHP diet compared with hypo-energetic CD diet, while achieving concurrent body weight loss of 5-7 percent in both groups. Levels of HbA1c will be measured at baseline, week 2, 4, 5 and 6. HbA1c will be expressed in mmol/mol.

SECONDARY OUTCOMES:
Change in hepatic fat content after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  Hepatic fat content will be assessed by magnetic resonance spectroscopy (MRs) at baseline and week 6.
Change in fasting plasma triglycerides during 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  Levels of triglycerides will be measured from fasting at baseline, week 2, 4, 5 and 6. Triglycerides will be expressed in mmol/L.

OTHER OUTCOMES:
Change in fat content subcutaneously, viscerally and ectopically in pancreas and skeletal muscle after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  Subcutaneous, visceral and ectopic fat in pancreas and skeletal muscle will be assessed by magnetic resonance imaging/spectroscopy (MRi/s) at baseline and week 6.
Change in lean body mass (LBM) after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  LBM will be assessed by dual-energy X-ray absorptiometry (DXA) at baseline and week 6. Changes will be expressed in kilograms (kg).
Change in fat mass (FM) after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  FM will be assessed by dual-energy X-ray absorptiometry (DXA) at baseline and week 6. Changes will be expressed in kilograms (kg).
Change in diurnal blood pressure (DBP) after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  DBP will be assessed over 24 hours by a blood pressure monitor (Ontrak 90227 from Spacelabs Healthcare) at baseline and week 6. DBP will be expressed in mmHg.
Change in heart rate variability (HRV) after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  HRV will be assessed by 48-hour Holter-monitoring (Faros 360 from Bittium) at baseline and week 6.
Change in diurnal glycemia after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  Glycemia will be assessed using 7-day continuous glucose monitoring (CGM) (FreeStyle Libre Pro from Abbott) at baseline and week 6.
Change in glycemic variability after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  Glycemic variability will be assessed using 7-day continuous glucose monitoring (CGM) (FreeStyle Libre Pro from Abbott) at baseline and week 6.
Change in insulin sensitivity after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  Insulin sensitivity will be assessed based on a 4-hour oral glucose tolerance test (OGTT) at baseline and week 6 and expressed by the Matsuda Index.
Change in beta-cell function after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  Beta-cell function will be assessed based on a 4-hour oral glucose tolerance test (OGTT) at baseline and week 6 and expressed by the Insulinogenic Index and Disposition Index.
Change in Homeostasis Model Assessment (HOMA) of insulin resistance and beta-cell function after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  HOMA will be performed at baseline and week 6 and expressed by HOMA-IR and HOMA-beta.
Change in lipid profile after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  Lipid profile, including lipoproteins will be assessed from fasting at baseline and week 6.
Change in glucose after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  Glucose will be measured during a 4-hour oral glucose tolerance test (OGTT) at baseline and week 6. Glucose will be expressed in mmol/L.
Change in insulin after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  Insulin will be measured during a 4-hour oral glucose tolerance test (OGTT) at baseline and week 6. Insulin will be expressed in pmol/L.
Change in C-peptide after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  C-peptide will be measured during a 4-hour oral glucose tolerance test (OGTT) at baseline and week 6. C-peptide will be expressed in pmol/L.
Change in non-esterified fatty acids (NEFA) after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  NEFA metabolism will be assessed using the minimal model technique based on an oral glucose tolerance test (OGTT) at baseline and week 6. NEFA will be expressed in micromol/L.
Change in triglycerides after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  Triglycerides will be measured during a 4-hour oral glucose tolerance test (OGTT) at baseline and week 6. Triglycerides will be expressed in mmol/L.
Change in glucagon after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  Glucagon will be measured during a 4-hour oral glucose tolerance test (OGTT) at baseline and week 6. Glucagon will be expressed in pmol/L.
Change in glucagon-like-peptide-1 (GLP-1) after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  GLP-1 will be measured during a 4-hour oral glucose tolerance test (OGTT) at baseline and week 6. GLP-1 will be expressed in pmol/L.
Change in glucose-dependent insulinotropic polypeptide (GIP) after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  GIP will be measured during a 4-hour oral glucose tolerance test (OGTT) at baseline and week 6. GIP will be expressed in pmol/L.
Change in peptide YY (PYY) after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  PYY will be measured during a 4-hour oral glucose tolerance test (OGTT) at baseline and week 6. PYY will be expressed in pmol/L.
Change in ghrelin after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  Ghrelin will be measured during a 4-hour oral glucose tolerance test (OGTT) at baseline and week 6. Ghrelin will be expressed in pmol/L.
Change in cholecystokinin (CCK) after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  CCK will be measured during a 4-hour oral glucose tolerance test (OGTT) at baseline and week 6. CCK will be expressed in pmol/L.
Change in gastrin after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  Gastrin will be measured during a 4-hour oral glucose tolerance test (OGTT) at baseline and week 6. Gastrin will be expressed in pmol/L.
Change in growth hormone (GH) after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  GH will be measured during a 4-hour oral glucose tolerance test (OGTT) at baseline and week 6. GH will be expressed in ng/mL.
Change in insulin-like growth factor-1 (IGF-1) after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  IGF-1 will be measured from fasting at baseline and week 6. IGF-1 will be expressed in ng/mL.
Change in insulin-like growth factor-binding protein 1 (IGFBP-1) after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  IGFBP-1 will be measured during a 4-hour oral glucose tolerance test (OGTT) at baseline and week 6. IGFBP-1 will be expressed in ng/mL.
Change in leptin after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  Leptin will be measured from fasting at baseline and week 6. Leptin will be expressed in ng/mL.
Change in adiponectin after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  Adiponectin will be measured from fasting at baseline and week 6. Adiponectin will be expressed in microg/mL.
Change in tumor necrosis factor alpha (TNF-alpha) after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  TNF-alpha will be measured from fasting at baseline and week 6 and expressed in pg/mL.
Change in interleukin-6 (IL-6) after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  IL-6 will be measured from fasting at baseline and week 6 and expressed in pg/mL.
Change in high-sensitive C-reactive protein (hsCRP) after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  hsCRP will be measured from fasting at baseline and week 6 and expressed in mg/L.
Change in renal function assessed from eGFR and diurnal excretion of albumin after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  eGFR and diurnal excretion of albumin will be assessed at baseline and week 6.
Change in urinary excretion of urea and glucose after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  Urinary excretion of urea and glucose will be assessed at baseline and week 6.
Change in urinary oxidative DNA and RNA modifications after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  Urinary oxidative DNA and RNA modifications will be assessed at baseline and week 6.
Change in subjective satiety after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  Subjective satiety will be assessed by a self-reported visual analog scale (VAS) questionnaire with four questions regarding experienced satiety (range 0-100 mm) integrated into one composite satiety score at baseline and week 6.
Change in health-related quality of life (HRQoL) after 6 weeks of hypo-energetic CRHP diet compared with hypo-energetic CD diet. | 6 weeks
  HRQoL will be assessed using a self-reported 36-item Short-Form (SF-36) health survey with 36 questions regarding different domains of HRQoL (each scoring from 0-100 points) at baseline and week 6. HRQoL will be reported as composite scores; a physical and mental component summary (PCS/MCS) score.

CONTACTS AND LOCATIONS:
Overall Officials: Steen B Haugaard, Professor, Principal Investigator — Dept. of Endocrinology, Copenhagen University Hospital Bispebjerg
Locations (1):
- Bispebjerg Hospital, Copenhagen, Copenhagen NV, Denmark

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) may be shared by request to the corresponding author in accordance with the Danish Data Protection Agency.

REFERENCES:
- [Derived] Thomsen MN, Skytte MJ, Samkani A, Weber P, Fenger M, Frystyk J, Hansen E, Holst JJ, Madsbad S, Magkos F, Thomsen HS, Walzem RL, Haugaard SB, Krarup T. Replacing dietary carbohydrate with protein and fat improves lipoprotein subclass profile and liver fat in type 2 diabetes independent of body weight: evidence from 2 randomized controlled trials. Am J Clin Nutr. 2025 Feb;121(2):224-231. doi: 10.1016/j.ajcnut.2024.11.030. Epub 2024 Nov 29. PMID 39617302
- [Derived] Jensen NJ, Wodschow HZ, Skytte MJ, Samkani A, Astrup A, Frystyk J, Hartmann B, Holst JJ, Larsen TM, Madsbad S, Magkos F, Miskowiak KW, Haugaard SB, Krarup T, Rungby J, Thomsen MN. Weight-loss induced by carbohydrate restriction does not negatively affect health-related quality of life and cognition in people with type 2 diabetes: A randomised controlled trial. Clin Nutr. 2022 Jul;41(7):1605-1612. doi: 10.1016/j.clnu.2022.05.005. Epub 2022 May 18. PMID 35679680
- [Derived] Thomsen MN, Skytte MJ, Samkani A, Carl MH, Weber P, Astrup A, Chabanova E, Fenger M, Frystyk J, Hartmann B, Holst JJ, Larsen TM, Madsbad S, Magkos F, Thomsen HS, Haugaard SB, Krarup T. Dietary carbohydrate restriction augments weight loss-induced improvements in glycaemic control and liver fat in individuals with type 2 diabetes: a randomised controlled trial. Diabetologia. 2022 Mar;65(3):506-517. doi: 10.1007/s00125-021-05628-8. Epub 2022 Jan 7. PMID 34993571